CLINICAL TRIAL: NCT02464826
Title: A Pilot Study - Safety and Efficacy of Nailprotex® for Onychomycosis Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Efficacynailprotex
Record Dates: First submitted 2015-04-30; First posted 2015-06-08 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Onychomycosis; Chronic Paronychia
Keywords: Onychomycosis; Chronic paronychia; Treatment
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Edit arms (Experimental): Nailprotex apply to the abnormal nail twice daily
  Interventions: Drug: Nailprotex

INTERVENTIONS:
Drug: Nailprotex — Nailprotex apply to the abnormal nail twice daily

SUMMARY:
This study was designed to demonstrate the efficacy of this product in non-dermatophyte (Scytalidium dimidiatum) onychomycosis and chronic paronychia treatment in Thai patients.

DETAILED DESCRIPTION:
Onychomycosis is the common superficial fungal skin infection in general population. According to the previous study, the prevalence of tinea pedis and onychomycosis in general Thai population were 3.8% and 1.7% respectively. However, this problem has been neglected for treatment due to asymptomatic clinical manifestations and low effects in quality of life.

In Thailand, the previous studies reported that the aetiological pathogens of this disorder were non-dermatophyte mold (51.6%), dermatophyte (36.3%) and yeast (6%). Additionally, Scytalidium dimidiatum was the majority causative agents in non-dermatophyte mold.

Systemic therapy such as azoles group and terbinafine is recommended for the standard management of tinea capitis. In contrast, a prolonged course may be induce serious side effects. So that topical therapy is the alternative treatment in older patients who are limited in drug usage. Especially, non-dermatophyte onychomycosis is the recalcitrant condition. Moreover, none of the standard regimen is recommended.

Nailprotex® is the novel topical treatment in onychomycosis and chronic paronychia. The active ingredient is phenol which is extracted from Olea European leaf. It is able to inhibit the fungal growth. Additionally, this product has been applied for nail care in many European countries over 10 years. The serious side effects have never been reported. Therefore, this study was designed to demonstrate the efficacy of this product in non-dermatophyte (Scytalidium dimidiatum) onychomycosis and chronic paronychia treatment in Thai patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants was 18 years old or above.
* Participants were diagnosed Scytalidium dimidiatum onychomycosis or chronic paronychia by dermatologists based on clinical presentation and mycological identification.
* Participants accept the aim of this project and sign the consent form by themselves.

Exclusion Criteria:

* Participants have other nail disorders before participate the research.
* Participants have the history of immunocompromised host.
* Participants were diagnosed onychomycosis more than 3 nails or matrix involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The change in the severity of onychomycosis by using SCIO (Scoring Clinical Index for Onychomycosis) score from baseline and 6 months-after using Nailprotex® | 6 months
  Patients who were treated by Nailprotex® in this study were evaluated the severity of onychomycosis by using SCIO (Scoring Clinical Index for Onychomycosis) score at baseline and after using Nailprotex® 6 months. Then the change in SCIO score was analyzed in percentage and compare mean.

SECONDARY OUTCOMES:
The side effects of Nailprotex® | 6 months
  The side effects of Nailprotex® was observed in patients from date of first application or first side effects documented progression until the date of end of study, assessed up to 6 months.
Mycological cure rate which mean KOH and fungal culture result are both nagative after using Nailprotex® at 6 month after treated with Nailprotex® | 6 months
  Patients who were treated by Nailprotex® in this study were evaluated the results of laboratory investigation (KOH examination and fungal culture) at baseline and after using Nailprotex® 6 months. Then mycological cure rate was analyzed in percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Charussri - Leeyaphan, MD., Principal Investigator — Department of Dermatology Faculty of Medicine, Siriraj Hospital Mahidol University
Locations (1):
- Department of Dermatology Siriraj Hospital, Bangkoknoi, Bangkok, Thailand